CLINICAL TRIAL: NCT04436211
Title: A Prospective Randomized Controlled Trial Evaluating Patient Specific Total Knee Arthroplasty Using Kinematic Alignment Versus Ligament-balanced, Mechanical Alignment
Brief Title: Kinematic- Versus Ligament-balanced Mechanical Alignment in TKA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 032020
Record Dates: First submitted 2020-04-01; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Osteo Arthritis Knee
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TKA (mechanical alignment)
  Interventions: Procedure: Total Knee Arthroplasty
- TKA (kinematic alignment)
  Interventions: Procedure: Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — The common procedure of Total Knee Arthroplasty is investigated in order to compare the techniques of implantation (kinematic vs mechanical alignment)

SUMMARY:
A promising new approach in total knee arthroplasty (TKA) for severe osteoarthritis of the knee joint is the the kinematic aligned procedure (KA). This technique provides prosthesis-positioning based on natural and individual axes of movement.

Although first series have shown satisfying results, further verification by prospective studies and final meta-analyses will be required.

Thus, the kinematic alignment represents one of the few new developments in TKA.

Provided that patients are willing to participate in the study, patients data are collected preoperatively and during routine follow-up examinations and evaluated prospectively. Patients will receive either a conventionally mechanical aligned arthroplasty or a kinematical aligned TKA, according to a randomized procedure.

The kinematic alignment will be achieved by the use of custom-made cutting-blocks. Therefore, the patients will undergo a computed tomography of the whole leg on the affected side. This is mandatory in order to provide the individually produced cutting blocks.

In order to ensure comparability, patients are stratified regarding their age and gender before inclusion.

Outcome will be measured by the use of standard scoring systems regarding function, pain and ROM (range of motion) three, six and 12 months after surgery.

This study is a monocentric, prospective, randomized and controlled open study.

ELIGIBILITY:
Inclusion Criteria:

- Severe osteoarthritis of the knee joint, intended for total knee arthroplasty

Exclusion Criteria:

- malalignment with varus of more than 5° or valgus malpositioning, joint instability

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case control study of 50 patients receiving a kinematical aligned TKA and 50 patients receiving a mechanical aligned TKA.
  In order to ensure comparability, patients are stratified regarding their age and gender before inclusion
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-02-15 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Change of Range of Motion (ROM) after kinematic vs mechanical aligned TKA | 3; 6; 12 months
  To assess range of motion a Standard Goniometer will be used. Measurements will be obtained after 3, 6, 12 months
Change of Pain after kinematic vs mechanical aligned TKA | 3; 6; 12 months
  The pain will be measured with the Visual Analog Scale (VAS), ranging from 1 to 10. 1 is meaning no pain, 10 is meaning the worst pain imaginable.
Change of Function after kinematic vs mechanical aligned TKA (OKS) | 3; 6; 12 months
  Function of the artificial joint will be assessed by the use of the Oxford Knee Score (OKS). The OKS is a patient reported outcome measure that consists of 12 questions about an individual's activities of daily living and how they have been affected by pain after total knee arthroplasty. All questions are scored from 0-4 where four is the best outcome and total scores range from 0 (worst outcome) to 48 (best outcome).
Change of Function after kinematic vs mechanical aligned TKA (WOMAC) | 3; 6; 12 months
  Function of the artificial joint will be assessed by the use of the Western Ontario and McMaster Universities Arthritis Index Score (WOMAC). The WOMAC survey is comprised of 24 items divided into three subscales: Pain (5 items), stiffness (2 items), and physical function (17 items). Patients are asked a range of questions about their ability to carry out daily activities such as using the stairs, rising from sitting, lying in bed and conducting light or heavy domestic duties. All the items are scored on a scale of 0-4 (lower scores indicate lower levels of symptoms or physical disability). Values are summed up for a combined WOMAC score.
Change of Function after kinematic vs mechanical aligned TKA (KSS) | 3; 6; 12 months
  Function of the artificial joint will be assessed by the use of the Combined Knee Society Score (KSS). The KSS has a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria